CLINICAL TRIAL: NCT03885856
Title: Clinical & Radiological Assessment of Rotator Cuff Healing After Single Row Vs. Double Row Rotator Cuff Repair; a Comparative Study
Brief Title: Clinical & Radiological Assessment of Rotator Cuff Healing After Single Row Vs. Double Row Rotator Cuff Repair
Acronym: RCR
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00339; ch19Taha
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Rotator Cuff Injury
Keywords: rotator cuff repair; rotator cuff tear; single row repair technique; double row repair technique
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- single row repair technique: patients surgically treated for rotator cuff lesion by single row repair technique
  Interventions: Other: single row repair technique
- double row repair technique: patients surgically treated for rotator cuff lesion by double row repair technique
  Interventions: Other: double row repair technique

INTERVENTIONS:
Other: single row repair technique — single row repair technique
  Groups: single row repair technique
Other: double row repair technique — double row repair technique
  Groups: double row repair technique

SUMMARY:
This study is to analyse whether there is a difference in clinical and radiological outcomes between single row and double row repair techniques for the treatment of shoulder's rotator cuff tears.

DETAILED DESCRIPTION:
A tear of the rotator cuff is one of the most common disorders of the shoulder and can have a significant effect on daily activities as a result of a loss of motion and strength. The goal of rotator cuff repair is to treat the patient's current clinical symptoms and improve shoulder function and to prevent the long-term consequences of rotator cuff arthropathy. This project aims at a retrospective analysis of preexisting risk factors for sustaining rotator cuff injury as well as for failing to reach the previous functional level, used surgical technique -either single row repair or double row repair- and its significance for the functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Treated by single row or double row repair technique for shoulder's rotator cuff tears
* Time lapse from injury to surgery ranges from one day to less than 1 year
* Availability of clinical and radiological outcomes from 6 months to 1 year follow up

Exclusion Criteria:

* Massive irreparable tear
* Patient has frozen shoulder
* Chronically retracted tendons and atrophic rotator cuff muscles

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for rotator cuff lesion either traumatic or degenerative at the University Hospital Basel and Kantonsspital BaselLand between 01.01.2015 and 30.1.2018
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Radiologic assessment of surgical treatment of rotator cuff tear | directly postoperative (within 24 hours after surgery)
  X-ray shoulder for assessment of acromiohumeral space and morphology (Millimeters)
Magnetic resonance imaging (MRI) of surgical treatment of rotator cuff tear | directly postoperative (within 24 hours after surgery)
  MRI shoulder to asses morphology of shoulder
Ultrasonography of surgical treatment of rotator cuff tear | From 6 months up to 1 year postoperative
  Ultrasonography to evaluate the healing of the tendon at the bone interface and degree of gap Formation (degree)

SECONDARY OUTCOMES:
Active range of motion | At six months and one year follow up after surgery
  Active range of motion of shoulder (degrees)
Passive range of motion | At six months and one year follow up after surgery
  Passive range of motion of shoulder (degrees)
Use of analgesics | At six months after surgery
  Use of analgesics (yes/no)
Use of analgesics | At one year follow up after surgery
  Use of analgesics (yes/no)

OTHER OUTCOMES:
Change in The American Shoulder and Elbow Surgeons Shoulder Score (ASES) | At six months and one year follow up after surgery
  The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. The patient questions focus on joint pain ( Visual Analogue Scale ranging from 0 = "no pain at all" to 10 = "pain as bad as it can be"), instability, and activities of daily living (ranging from "unable to do" to " not difficult"). The pain and functional portions are summed to obtain the final ASES score with higher scores indicating better outcomes.
Pain at rest (yes/no) | At six months after surgery
  Pain at rest (yes/no)
Change in Constant-Murley score (CMS) | At six months and one year follow up after surgery
  Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function
Pain at rest (yes/no) | At one year follow up after surgery
  Pain at rest (yes/no)
Pain under stress (yes/no) | At six months after surgery
  Pain under stress (yes/no)
Pain under stress (yes/no) | At one year follow up after surgery
  Pain under stress (yes/no)
Number of Reoperations (quantity) | Summarized over a one year follow up period after surgery
  Number of Reoperations (quantity)
Number of Rehospitalizations (quantity) | Summarized over a one year follow up period after surgery
  Number of Rehospitalizations (quantity)

CONTACTS AND LOCATIONS:
Overall Officials: Mohy Taha, Dr. med, Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics, Basel, Switzerland